CLINICAL TRIAL: NCT04282655
Title: The Effect of a Continuous Milk Warming System on Feeding Tolerance and Growth Rates in Very Low Birth Weight Infants
Brief Title: Effect of Milk Warming on the Very Low Birth Weight Infant
Acronym: VLBW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6748
Record Dates: First submitted 2019-01-09; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Very Low Birth Weight Infant; Weight Gain; Feeding Disorder Neonatal
Keywords: breast milk; milk warming
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Intervention Model Description: Randomized prospective quasi-experimental controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard method of warming breast milk in a hot water bath prior to feeding.
  Interventions: Other: Control
- Treatment Guardian Milk Warmer (Medela TM) (Experimental): External continuous milk warmer that heats milk within the tubing just posterior to the feeding tube to provide milk at body temperature for feeding infusion.
  Interventions: Other: Treatment Guardian Milk Warmer (Medela TM)

INTERVENTIONS:
Other: Treatment Guardian Milk Warmer (Medela TM) — Infants were randomized to receive prepared syringes of breast milk via the continuous milk warmer (treatment arm)
  Other Names: Continuous milk warmer (Guardian Warmer, Medela™)
  Arms: Treatment Guardian Milk Warmer (Medela TM)
Other: Control — Standard warming procedure of breast milk in syringe prior to feeding.
  Arms: Control

SUMMARY:
This study will compare if using a continuous milk warmer to warm breast milk compared to the standard method of warming breast milk in a hot water bath improves weight gain and feeding tolerance in infants born at 32 weeks gestation or less over a ten-day period. The standard method does not keep the breast milk at a consistent temperature during the feeding. A continuous milk warmer maintains the breast milk at body temperature throughout the feeding. It is unknown which method improves weight gain and feeding tolerance in very low birth weight infants.

DETAILED DESCRIPTION:
The aim of this randomized prospective quasi-experimental study is to determine if providing body temperature breast milk feedings to very low birth weight infants through use of continuous milk warmer improves feeding tolerance and weight gain compared to a standard milk warming technique.

Warming breast milk in a hot water bath just prior to feeding prior to feeding in the neonatal intensive care unit is a common practice. However, little evidence is available to support a standard warming method. This method allows inconsistent temperatures at time of feeding and progressive cooling of the milk during the feeding. No published study used a continuous warming device that delivered milk at a consistent physiological temperature throughout the feeding. The continuous warmer externally heats milk in the tubing just posterior to the feeding tube to provide body temperature milk to the infant.

A convenience sample from the Children's Hospital at OU Medical Center of 50 very low birth weight infants will be randomly assigned to either the experimental or control group for ten days. The experimental group will receive warmed feedings through the duration of the feeding through the use of the Guardian Warmer™, a continuous milk warming device. A control group will receive breast milk feedings warmed using the standard milk warming methods. Feeding tolerance and weight gain over the ten-day period will be used to evaluate the effectiveness of continuous milk warming.

ELIGIBILITY:
Inclusion Criteria:

• Gestational age 28-32 weeks on full enteral feeding of breast milk

Exclusion Criteria:

* Mechanical ventilation
* Positive End Expiratory Pressure (PEEP)
* Total parenteral nutrition, or any congenital anomalies
* Severe to moderate respiratory disease
* Previous medical or surgical necrotizing enterocolitis.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Weight Gain | At study completion, 10 days.
  Comparison of two groups for weight gain over time in grams
Feeding Intolerance | At study completion, 10 days
  Comparison of feeding tolerance between groups using a residual algorithm

SECONDARY OUTCOMES:
Head Circumference | At study completion, 10 days
  frontal-occipital circumference in centimeters
Body Length | At Study completion, 10 days
  Length as measured in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Kris Sekar, MD, Principal Investigator — OUHSC Dept of Pediatrics, Neonatal-Perinatal Medicine; Susan M Bedwell, DNP, Principal Investigator — Univeristy of Oklahoma, The Children's Hospital
Locations (1):
- University of Oklahoma, The Children's Hospital, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson CA, Berseth CL. Neither motor responses nor gastric emptying vary in response to formula temperature in preterm infants. Biol Neonate. 1996;70(5):265-70. doi: 10.1159/000244375. PMID 8955912
- [Background] Blumenthal I, Lealman GT, Shoesmith DR. Effect of feed temperature and phototherapy on gastric emptying in the neonate. Arch Dis Child. 1980 Jul;55(7):562-4. doi: 10.1136/adc.55.7.562. PMID 7436507
- [Background] Dumm M, Hamms M, Sutton J, Ryan-Wenger N. NICU breast milk warming practices and the physiological effects of breast milk feeding temperatures on preterm infants. Adv Neonatal Care. 2013 Aug;13(4):279-87. doi: 10.1097/ANC.0b013e31829d8c3a. PMID 23912021
- [Background] Eckburg JJ, Bell EF, Rios GR, Wilmoth PK. Effects of formula temperature on postprandial thermogenesis and body temperature of premature infants. J Pediatr. 1987 Oct;111(4):588-92. doi: 10.1016/s0022-3476(87)80127-0. PMID 3116191
- [Derived] Bedwell SM, Buster B, Sekar K. The Effect of a Continuous Milk Warming System on Weight Gain in Very Low Birth-Weight Infants: A Randomized Controlled Trial. Adv Neonatal Care. 2021 Aug 1;21(4):E86-E92. doi: 10.1097/ANC.0000000000000818. PMID 33427754